CLINICAL TRIAL: NCT04876898
Title: High Body Mass Index and Severity of Coronavirus Disease 2019 (Covid-19): a Cohort Study
Brief Title: High Body Mass Index and Severity of Coronavirus
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Gad Sayed Gad, ass.prof anesthesia department, South Valley University
Other Study IDs: BMI_COVID19
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prospective cohort in high body mass index patient with covid 19 — A cohort study included 114 adult patients with confirmed COVID-19 were categorized by BMI levels

SUMMARY:
A cohort study included 114 adult patients with confirmed COVID-19 were categorized by BMI levels on admission: overweight (25-29.9 kg/m2), and obesity (four categories: 30-34.9 kg/m2, 35-39.9 kg/m2, 40-44.9 kg/m2, and ≥45 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* confirmed COVUID 19 infection
* body mass index more than 25kg/m2

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 114 adult patients with confirmed COVID-19 were categorized by BMI levels on admission: overweight (25-29.9 kg/m2), and obesity (four categories: 30-34.9 kg/m2, 35-39.9 kg/m2, 40-44.9 kg/m2, and ≥45 kg/m2). Pneumonia, severe pneumonia, and ICU admission rate were our primary outcomes, complications, and length of hospital stay was the secondary outcome.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
pneumonia | 30 days
  patients percentages
sever pneumonia | 30 days
  patients percentages
ICU admission | 30 days
  patients percentages

SECONDARY OUTCOMES:
length of hospital stay | 30 days
  days
clinical complication | 30 days
  patients percentages

CONTACTS AND LOCATIONS:
Overall Officials: Gad S Gad, phd, Principal Investigator — ass prof ,anesthesia and ICU ,south valley university,Qena .Egypt
Locations (1):
- Gad sayed Gad, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No